CLINICAL TRIAL: NCT00870961
Title: Vitamin D Intervention For Colon Cancer Prevention In African-Americans-A Pilot Study
Brief Title: Vitamin D Supplement in Preventing Colon Cancer in African Americans With Colon Polyps
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI changed institutions and accrual was not completed.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NU 08I3; P30CA060553 (NIH); NU-08I3; STU00005964 (Other: Northwestern University IRB)
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer; Precancerous Condition
Keywords: colon cancer; rectal cancer; adenomatous polyp
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms; Adenomatous Polyps | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Experimental): Patients receive oral cholecalciferol (vitamin D3) supplementation daily for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: cholecalciferol
- Arm II (Placebo Comparator): Patients receive oral placebo supplementation daily for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of vitamin D may keep colorectal cancer from forming in patients with colon polyps.

PURPOSE: This randomized phase I trial is studying a vitamin D supplement to see how well it works compared with a placebo in preventing colorectal cancer in African Americans with colon polyps.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the accrual rate of African Americans with adenomatous polyps to a 6-month randomized intervention trial comprising supplementation with either cholecalciferol (vitamin D3) or placebo.
* To determine the compliance rates in patients treated with these regimens.

Secondary

* To compare changes in pre- and post-treatment vitamin D levels in patients treated with these regimens.
* To correlate vitamin D levels with vitamin D modifiers, such as levels of skin pigmentation, dietary vitamin D intake, and sun exposure in this patient population.

OUTLINE: Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral cholecalciferol (vitamin D3) supplementation daily for up to 6 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo supplementation daily for up to 6 months in the absence of disease progression or unacceptable toxicity.

Patients complete questionnaires about demographics, dietary vitamin D intake, personal history (e.g., ancestry, alcohol and tobacco intake, occupation, height, and weight), medical history (e.g., personal and family history of colorectal cancer and polyps), and ultraviolet radiation exposure.

Blood samples are collected at baseline and at 6 months for correlative laboratory studies. Blood samples are analyzed for vitamin D levels by enzyme immunoassay. Patients also undergo assessment of skin pigmentation in sunprotected and sunexposed areas of skin by reflectance spectrometry at baseline.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenomatous polyp

  * At least 1 adenoma
* Self-identified as an African American AND undergoing screening or diagnostic colonoscopy at the University of Chicago
* No history of colon or rectal cancer or hereditary or familial colon cancer (e.g., hereditary non-polyposis colon cancer or familial adenomatous polyposis)

PATIENT CHARACTERISTICS:

* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Albumin ≥ 3.0 mg/dL
* Baseline serum calcium level normal
* Not pregnant
* No history of thyroid disease
* No history of renal stones

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other concurrent vitamin D intake

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Rate of compliance as assessed at 6 months | Following 6 months of study treatment
Rate of accrual | After accrual goal is reached

SECONDARY OUTCOMES:
Changes in pre- and post-treatment vitamin D levels | At baseline and following completion of study treatment
Correlation of vitamin D levels with vitamin D modifiers (e.g., levels of skin pigmentation, dietary vitamin D intake, and sun exposure) | After completion of study treatment & final colonic biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Halla Nimeiri, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois